CLINICAL TRIAL: NCT03013699
Title: Improving Dietary Patterns in Head and Neck Cancer Survivors to Optimize Disease Outcomes and Supportive Care: A Pilot/Feasibility Intervention Study
Brief Title: Diet Intervention, Head and Neck Cancer, Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: X140813004
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Head and Neck Cancer
Keywords: diet; nutrition; survival; recurrence; cruciferous; dark leafy greens
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Dietary Care (Active Comparator): Participants receive standard educational materials that focus on healthy eating for cancer survivors and the opportunity to briefly discuss nutrition-related concerns with the Registered Dietitian weekly.
  Interventions: Behavioral: Usual Dietary Care
- Cruciferous and Dark Leafy Green Intervention (Experimental): Participants receive individual dietary counseling from a Registered Dietitian who will focus on increasing intake of cruciferous and green leafy vegetables while addressing any disease- and treatment-related eating difficulties experienced by the participant.
  Interventions: Behavioral: Cruciferous and Dark Leafy Green Intervention

INTERVENTIONS:
Behavioral: Cruciferous and Dark Leafy Green Intervention — Participants receive individual dietary counseling from a Registered Dietitian who will focus on increasing intake of cruciferous and green leafy vegetables while addressing any disease- and treatment-related eating difficulties experienced by the participant.
  Arms: Cruciferous and Dark Leafy Green Intervention
Behavioral: Usual Dietary Care — Participants receive standard educational materials that focus on healthy eating for cancer survivors and the opportunity to briefly discuss nutrition-related concerns with the Registered Dietitian weekly.
  Arms: Usual Dietary Care

SUMMARY:
This study will examine the effects of a dietary intervention in post-treatment head and neck cancer survivors on the ability to function physically, tiredness, and quality of life, as well as on changing markers in the blood that are associated with better recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible to participate if they are 1) diagnosed with Stage I - IV oral, hypopharyngeal, nasopharyngeal, oropharyngeal, or laryngeal cancer; 2) age 19+; 3) at least 6 months - 2 years post-treatment; 4) able to consume foods orally; 5) no evidence of disease; 6) English-speaking

Exclusion Criteria:

Patients will not be eligible to participate if they have 1) dementia or organic brain syndrome; 2) severe emotional distress; 3) active schizophrenia; 3) another diagnosis of cancer in the past five years (not including skin or cervical cancer in situ)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of patients excluded or not agreeing to participate | Baseline
  Feasibility measure
Adherence to study protocol activities (research records and diet intake self-report) | Throughout 12 week study period
  Feasibility measure (e.g., percent of assessments completed, percent of counseling phone calls completed, servings of cruciferous vegetables eaten, etc.)
Attrition rates | Throughout 12 week study period
  Feasibility measure
Adverse events with reporting according to institutional review board policy | Throughout 12 week study period
Questionnaire | At conclusion of 12 week study period
  Participant satisfaction
Questionnaire | At conclusion of 12 week study period
  Intervention preferences

SECONDARY OUTCOMES:
DNA methylation | At beginning and end of 12 week study period
Serum cytokines | At beginning and end of 12 week study period
Quality of life (assessed using the Functional Assessment of Cancer Therapy Head and Neck index) | At beginning and end of 12 week study period
Total energy and nutrient intakes | At beginning and end of 12 week study period
Covariates | At beginning of 12 week study period
  A questionnaire will collect a set of covariates used in the analyses (i.e., these do not represent individual outcomes; this is a group of covariates used in the data analyses). This group includes demographic characteristics (age, sex, race, ethnicity, education, income); lifestyle behaviors (tobacco use, alcohol consumption, exercise); medical history; cancer-specific clinical variables (tumor site, cancer stage, treatment modality); anthropometrics (height and weight)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Q. Rogers, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No